CLINICAL TRIAL: NCT06513507
Title: A Clinical Study to Assess the Efficacy of Cannabigerol in Patients with Active Rheumatoid Arthritis.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Raphael Pharma (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20441
Record Dates: First submitted 2024-07-17; First posted 2024-07-22 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Rheumatoid Arthritis; Inflammatory Disease
Keywords: Arthritis Treatment; Cannabinoid Therapy; Anti-CCP
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — cannabigerol

STUDY DESIGN:
Intervention Model Description: This is a single-group study with an exploratory longitudinal prospective design aimed at measuring the efficacy of purified cannabigerol (CBG) in patients with active rheumatoid arthritis.
Masking Description: No blinding will be performed in this study. All participants and investigators will know the treatment being administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CBG Treatment (Experimental): Participants will receive 0.5 milliliters of purified cannabigerol (CBG) in sesame oil once daily in the evening for a duration of eight weeks.
  Interventions: Dietary Supplement: Cannabigerol (CBG)

INTERVENTIONS:
Dietary Supplement: Cannabigerol (CBG) — The daily dose will consist of 50 mg of CBG. Blood tests will be conducted at Baseline, Week 2, Week 4, Week 6, and Week 8 to monitor inflammatory markers and immune response. Self-reported questionnaires will be completed at Baseline, Week 4, and Week 8 to assess symptoms and quality of life.

SUMMARY:
This is a single-group exploratory longitudinal prospective study lasting 8 weeks. The study aims to measure the efficacy of purified cannabigerol (CBG) in patients with active rheumatoid arthritis using laboratory and self-reported outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, over 25 years of age
* Positive anti-CCP blood test
* Active RA-related inflammation with at least 2 swollen joints
* University graduate
* Generally healthy with no uncontrolled chronic disease
* Able to read, understand, and sign informed consent
* Resides in the USA
* Willing to comply with study requirements and avoid other cannabis products during the study period

Exclusion Criteria:

* Pre-existing chronic conditions preventing adherence
* Severe allergic reactions requiring an Epi-pen
* Use of opiates in the last 4 weeks or cannabis in the last 8 weeks
* Pregnant or breastfeeding women
* Recent invasive medical procedure or surgery
* Active malignancy or ongoing oncology treatment
* Use of cytochrome P450 or 3A4 inhibitors
* History of substance abuse

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in inflammatory markers from Baseline to Week 8 | Baseline, Week 2, Week 4, Week 6, and Week 8
  Measurement of blood levels of ESR (Erythrocyte Sedimentation Rate), CRP (C-Reactive Protein), IL6 (Interleukin 6), and TNFa (Tumor Necrosis Factor-alpha) at Baseline, Week 2, Week 4, Week 6, and Week 8.

SECONDARY OUTCOMES:
Change in self-reported symptoms and quality of life from Baseline to Week 8 | Baseline, Week 4, and Week 8
  Evaluation of participant perceptions of the product's effect on symptoms of rheumatoid arthritis and quality of life using a study-specific questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Yes